CLINICAL TRIAL: NCT04603287
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of SI-B001, an EGFR/HER3 Bispecific Antibody, in Locally Advanced or Metastatic Epithelial Tumors
Brief Title: A Study of SI-B001, an EGFR/HER3 Bispecific Antibody, in Locally Advanced or Metastatic Epithelial Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001/CC-E/H3101
Record Dates: First submitted 2020-10-08; First posted 2020-10-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Epithelial Tumor
Keywords: Non-small cell lung cancer (NSCLC); Head and neck squamous cell carcinoma (HNSCC); Esophageal cancer; Colorectal cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive SI-B001 as intravenous infusion for the first cycle (4 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: SI-B001

INTERVENTIONS:
Drug: SI-B001 — Administration by intravenous infusion.

SUMMARY:
In phase Ia study, the safety and tolerability of SI-B001 in patients with locally advanced or metastatic epithelial malignancies will be investigated to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) of SI-B001.

In the phase Ib study, the safety and tolerability of SI-B001 at the phase Ia recommended dose will be further investigated, and recommended phase II dose (RP2D) for phase II clinical studies will be determined.

In addition, the preliminary efficacy, pharmacokinetic characteristics, and immunogenicity of SI-B001 in patients with locally advanced or metastatic epithelial tumors will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign the informed consent form voluntarily and follow the plan requirements.
2. No gender limit.
3. Age: ≥18 years old and ≤75 years old (stage Ia); ≥18 years old (stage Ib).
4. Expected survival time ≥ 3 months.
5. Locally advanced or metastatic epithelial malignancies are confirmed by histopathology and/or cytology that are incurable or currently without standard treatment.
6. Participants must agree to provide archived tumor tissue specimens or fresh tissue samples within 6 months of the primary tumor or metastasis; in phase Ia, if the participant is unable to provide tumor tissue samples, the investigator will evaluate whether the participant could be enrolled if other criteria are fit to join the group.
7. Participants must have at least one measurable lesion that meets the definition of RECIST v1.1.
8. Physical fitness score ECOG 0 or 1 point.
9. The toxicity of previous anti-tumor treatments has been restored to NCI-CTCAE v5.0 definition ≤ 1 (except for hair loss).
10. No serious cardiac dysfunction, left ventricular ejection fraction (LVEF) ≥50%, (hypersensitivity) troponin T<ULN.
11. The organ function must meet the following requirements and standards: a) Bone marrow function: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90 g/L; B) Liver function: total bilirubin (TBIL≤1.5 ULN), AST and ALT ≤2.5 ULN for participants without liver metastasis, AST and ALT ≤5.0 ULN for liver metastases; c) Kidney function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to the Cockcroft and Gault formula).
12. Coagulation function: International normalized ratio (INR)≤1.5×ULN, and activated partial thromboplastin time (APTT)≤1.5ULN.
13. Urine protein≤2%2B (measured with test paper) or≤1000mg/24h (urine).
14. For premenopausal women with childbearing potential, a pregnancy test must be taken within 7 days prior to the start of treatment. Serum or urine pregnancy must be negative and must be non-lactating; all participants (regardless of male or female) in the group should be treated throughout the treatment. Adequate barrier contraceptive measures should be taken during the treatment and 6 months after the treatment.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, major surgery, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other anti-tumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration; oral fluorouracil-like drugs such as S-1, capecitabine, or palliative radiotherapy within 2weeks prior to the first administration.
2. If there is a history of vaccination within 3 months prior to the first administration, it is allowed to receive inactivated influenza vaccine within 30 days prior to the first administration, and the treatment of live attenuated vaccine is not allowed.
3. Participants with history of severe heart disease, such as: symptomatic congestive heart failure (CHF) ≥ grade 2 (CTCAE 5.0), New York Heart Association (NYHA) ≥ grade 2 heart failure, history of transmural myocardial infarction, unstable angina pectoris etc.
4. Participants with prolonged QT interval (male QTc> 450 msec or female QTc> 470 msec), complete left bundle branch block, III grade atrioventricular block.
5. Active autoimmune diseases and inflammatory diseases, such as: systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., except for type I diabetes, hypothyroidism that can be controlled only by alternative treatment, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis).
6. Other malignant tumors were diagnosed within 5 years prior to the first administration with the following exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after radical resection.
7. Participants with poorly controlled hypertension by two kinds of antihypertensive drugs (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg).
8. Participants have grade 3 lung disease defined according to NCI-CTCAE v5.0, including participants with resting dyspnea, or requiring continuous oxygen therapy, or a history of interstitial lung disease (ILD).
9. Symptoms of active central nervous system metastasis. However, participants with stable brain metastasis or stable epidural spinal cord compression history can be included. Stable is defined as: a. With or without antiepileptic drugs, the seizure-free state lasts for more than 12 weeks; b. There is no need to use glucocorticoids; c. Continuous multiple MRI (scanning interval at least 8 weeks) showed a stable state in imaging.
10. Participants who have a history of allergies to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of SI-B001.
11. Participants have a history of autologous or allogeneic stem cell transplantation.
12. In the adjuvant (or neoadjuvant) treatment of anthracyclines, the cumulative dose of anthracyclines is> 360 mg/m2.
13. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number> 104) or hepatitis C virus (HCV) infection.
14. Participants with active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
15. Other conditions that the investigator believes that it is not suitable for participating in this clinical trial.
16. Participated in another clinical trial within 4 weeks prior to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 28 days after the first dose of SI-B001
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle (28 days) and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 28 days after the first dose of SI-B001
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle (within 28 days of the first administration).
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 28 days after the first dose of SI-B001
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of SI-B001.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of SI-B001. The type, frequency and severity of TEAE will be evaluated during the treatment of SI-B001.
Cmax | Up to 28 days after the first dose of SI-B001
  Maximum serum concentration (Cmax) of SI-B001 will be investigated.
Tmax | Up to 28 days after the first dose of SI-B001
  Time to maximum serum concentration (Tmax) of SI-B001 will be investigated.
T1/2 | Up to 28 days after the first dose of SI-B001
  Half-life (T1/2) of SI-B001 will be investigated.
AUC0-t | Up to 28 days after the first dose of SI-B001
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to 28 days after the first dose of SI-B001
  CL in the serum of SI-B001 per unit of time will be investigated.
Ctrough | Up to 28 days after the first dose of SI-B001
  Ctough is defined as the lowest serum concentration of SI-B001 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Incidence and titer of ADA of SI-B001 will be evaluated.
Nab (neutralizing antibody) | Up to approximately 24 months
  Incidence and titer of Nab of SI-B001 will be evaluated.
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of SI-B001 to the first date of either disease progression or death, whichever occurs first.
Overall survival | Up to approximately 24 months
  The OS is defined as the time from the participant's first dose of SI-B001 to the time of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang